CLINICAL TRIAL: NCT02172781
Title: A Double-blind, Randomised, Two-way Cross-over Study to Investigate the Pharmacokinetic and Pharmacodynamic Effects of a Single Additional Dose of 500 µg Ipratropium Bromide Unit Dose Vial Inhaled Via Nebuliser Versus Placebo After 19 Days of Treatment With Tiotropium Inhalation Capsules 18 µg q.d. in Male Healthy Volunteers.
Brief Title: Comparative Pharmacokinetics and Pharmacodynamics of Tiotropium With Ipratropium or Placebo After 19 Days of Tiotropium Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.239
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (5):
- Ipratropium - unit dose vial (Experimental)
  Interventions: Drug: Ipratropium - unit dose vial; Drug: Placebo matching ipratropium
- Tiotropium - inhalation capsule - low dose (Experimental)
  Interventions: Drug: Ipratropium - unit dose vial; Drug: Tiotropium - inhalation capsule; Drug: Placebo matching tiotropium; Drug: Placebo matching ipratropium
- Placebo matching tiotropium - inhalation capsule (Placebo Comparator)
  Interventions: Drug: Ipratropium - unit dose vial; Drug: Tiotropium - inhalation capsule; Drug: Placebo matching tiotropium; Drug: Placebo matching ipratropium
- Placebo matching to ipratropium - unit dose vial (Placebo Comparator)
  Interventions: Drug: Ipratropium - unit dose vial; Drug: Tiotropium - inhalation capsule; Drug: Placebo matching tiotropium; Drug: Placebo matching ipratropium
- Tiotropium - inhalation capsule - high dose (Experimental)
  Interventions: Drug: Ipratropium - unit dose vial; Drug: Tiotropium - inhalation capsule; Drug: Placebo matching ipratropium

INTERVENTIONS:
Drug: Ipratropium - unit dose vial
Drug: Tiotropium - inhalation capsule
  Arms: Placebo matching tiotropium - inhalation capsule; Placebo matching to ipratropium - unit dose vial; Tiotropium - inhalation capsule - high dose; Tiotropium - inhalation capsule - low dose
Drug: Placebo matching tiotropium
  Arms: Placebo matching tiotropium - inhalation capsule; Placebo matching to ipratropium - unit dose vial; Tiotropium - inhalation capsule - low dose
Drug: Placebo matching ipratropium

SUMMARY:
Comparative Pharmacokinetics and Pharmacodynamics of Tiotropium With Ipratropium or Placebo After 19 Days of Tiotropium Treatment

ELIGIBILITY:
Inclusion Criteria:

All participants in the study should be healthy males, ranging from 40 to 65 years of age and within ±20% of their normal weight (Broca-Index)

Each subject will have his medical history taken and will receive a complete medical examination (including blood pressure and pulse rate measurements) as well as a 12-lead ECG.

Haematological, hepatic and renal function tests will be carried out in the laboratory (Bioscentia GmbH, FRG). The subjects will fast for 8 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first drug administration.

In accordance with Good Clinical Practice (GCP) and local legislation all subjects will have given their written informed consent prior to admission to the study.

Following inclusion criteria were of special interest for this study:

* Normal spirometry as evidenced by a baseline FEV1 ≥ 80% of predicted normal value for age, height and sex. Predicted normal values will be calculated according to European Community of Coal and Steel (ECCS)
* Ability to perform technically satisfactory pulmonary function tests.

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders.
* History of orthostatic hypotension, fainting spells or blackouts.
* Chronic or relevant acute infections.
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator.
* Intake of drugs with a long half-life (≥ 24hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study.
* Use of any drugs which might influence the results of the trial up to seven days prior to enrolment in the study or during the study, among these all non-selective beta blockers, oral beta adrenergics or long-acting beta-adrenergics such as salmeterol and formoterol, and anticholinergic drugs including ATROVENT ®(ipratropium) by oral inhalation and ATROVENT® Nasal Spray.
* Participation in another trial with an investigational drug (≤ two months prior to administration or during trial).
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days.
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation (≥ 100 ml within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range.
* Excessive physical activities (within the last week before and during the study)

Following exclusion criteria are of special interest for the study:

* Subjects with known hypersensitivity to anticholinergic drugs.
* Subjects with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Subjects with known narrow-angle glaucoma

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2001-01; Primary Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
AUC - Area under the curve of the log-transformed value of salivary secretion after application of randomised treatment | over the interval from two hours to six hours on study day 19 and 22

SECONDARY OUTCOMES:
Cmax (Peak (maximum) plasma concentration) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
Cmax,ss (maximum observed concentration of the analyte in plasma at steady state) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
Tmax (time to reach the peak plasma concentration) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
Tmax, ss (Time to reach maximum concentration of the analyte in plasma at steady state) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
Cpre (predose concentration of the analyte in plasma) -Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
Cpre,ss (predose concentration of the analyte in plasma at steady state) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
AUC (area under the concentration time curve of the analyte in plasma) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
AUC,ss (area under the concentration time curve of the analyte in plasma at steady state) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
Ae (amount of analyte that is eliminated in urine) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
CLR (renal clearance of the analyte) - Tiotropium | Day1, day 7, day 19, day 22 ( before and different time points after dosing), day 2, day 3, day 20 (before dosing)
Cmax (Peak (maximum) plasma concentration) - Ipratropium | Day A1, A4 (before and after inhalation of ipratropium), day 19, day 22 (before, at end of ipratropium inhalation and different time points after tiotropium dosing), day 20 (10 min.before tiotropium dosing)
Tmax (time to reach the peak plasma concentration) - Ipratropium | Day A1, A4 (before and after inhalation of ipratropium), day 19, day 22 (before, at end of ipratropium inhalation and different time points after tiotropium dosing), day 20 (10 min.before tiotropium dosing)
AUC (area under the concentration time curve of the analyte in plasma) - Ipratropium | Day A1, A4 (before and after inhalation of ipratropium), day 19, day 22 (before, at end of ipratropium inhalation and different time points after tiotropium dosing), day 20 (10 min.before tiotropium dosing)
Ae (amount of analyte that is eliminated in urine) - Ipratropium | Day A1, A4 (before and after inhalation of ipratropium), day 19, day 22 (before, at end of ipratropium inhalation and different time points after tiotropium dosing), day 20 (10 min.before tiotropium dosing)
CLR (renal clearance of the analyte) - Ipratropium | Day A1, A4 (before and after inhalation of ipratropium), day 19, day 22 (before, at end of ipratropium inhalation and different time points after tiotropium dosing), day 20 (10 min.before tiotropium dosing)
Amount of Salivary secretion | Screening, A1, A4 ( before and after dosing of ipratropium), different time points at day 1, day 2, day 7, day 19 and 22 (before and after dosing of tiotropium and Ipratropium), day 20, day 23
FEV1 (Forced expiratory volume in one second) | Screening, A1, A4 ( before and after dosing of ipratropium), different time points at day 1, day 2, day 7, day 19 and 22 (before and after dosing of tiotropium and Ipratropium), day 20, day 23
FVC (Forced vital capacity) | Screening, A1, A4 ( before and after dosing of ipratropium), different time points at day 1, day 2, day 7, day 19 and 22 (before and after dosing of tiotropium and Ipratropium), day 20, day 23
MMEF25-75% (maximal mid-expiratory flow) | Screening, A1, A4 ( before and after dosing of ipratropium), different time points at day 1, day 2, day 7, day 19 and 22 (before and after dosing of tiotropium and Ipratropium), day 20, day 23
PEFR (peak expiratory flow rate) | Screening, A1, A4 ( before and after dosing of ipratropium), different time points at day 1, day 2, day 7, day 19 and 22 (before and after dosing of tiotropium and Ipratropium), day 20, day 23
Occurence of adverse events | Screening, A1-A6, B1-B23, end of study (within 8 days after last dosing tiotropium)